CLINICAL TRIAL: NCT03230370
Title: Does the Enhanced Rehabilitation Programs Facilitate the Motor Recovery After Stroke? A Multicenter Randomized Controlled Study (TIARAS Trial)
Brief Title: Does the Enhanced Rehabilitation Programs Facilitate the Motor Recovery After Stroke?
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No adequate funding
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Principal Investigator, Yen-Nung Lin, Director of Rehabilitation Department of Taipei Medical University WanFang Hospital, Taipei Medical University WanFang Hospital
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: N201705071
Record Dates: First submitted 2017-07-20; First posted 2017-07-26 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-09

CONDITIONS: Poststroke/CVA Hemiparesis
Keywords: intensity; rehabilitation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- enhanced upper-extremity program, EUEP (Experimental): Both groups receive routine rehabilitation including daily 50 mins of physical therapy and 50 mins of occupational therapy.
  The EUP group receives additional daily 50 mins program focusing on training of the hemiplegic upper extremity.
  The participants receive 20-day training over a 4-weekperiod. The additional program is designed to be specific to either upper-extremity or lower-extremity.
  Accordingly, one group can be used as the control group of the other one.
  Interventions: Other: UFT
- enhanced lower-extremity program,ELLP) (Experimental): Both groups receive routine rehabilitation including daily 50 mins of physical therapy and 50 mins of occupational therapy.
  The ELP group receives additional daily 50 mins program focusing on training of the hemiplegic lower extremity.
  The participants receive 20-day training over a4-weekperiod. The additional program is designed to be specific to either upper-extremity or lower-extremity.
  Accordingly,one group can be used as the control group of the other one.
  Interventions: Other: LFT

INTERVENTIONS:
Other: UFT — The EUEP group receives additional daily 50 mins program focusing on training of the hemiplegic upper extremity,
  Arms: enhanced upper-extremity program, EUEP
Other: LFT — The ELEP group receives additional daily 50 mins program focusing on training of the hemiplegic lower extremity.
  Arms: enhanced lower-extremity program,ELLP)

SUMMARY:
Study purpose This study will explore whether an additional rehabilitation program that focus on either upper or lower extremity training facilitate the recovery in upper or lower extremity.

The recovery in both neurological status and motor functions will be explored.

DETAILED DESCRIPTION:
Design A single-blinded (assessor-blinded) randomized controlled trial. Interventions The participants will be randomly assigned into two experiment groups (enhanced upper extremity program; and enhanced lower-extremity program).

Both groups receive routine rehabilitation including daily 50 mins of physical therapy and 50 mins of occupational therapy.

The enhanced upper extremity program group receives additional daily 50 mins program focusing on training of the hemiplegic upper extremity, while the enhanced lower-extremity program group receives additional daily 50 mins program focusing on training of the hemiplegic lower extremity. The participants receive 20-day training over a 4-week period. The additional program is designed to be specific to either upper-extremity or lower-extremity. Accordingly, one group can be used as the control group of the other one.

ELIGIBILITY:
Inclusion Criteria:

1. First-ever stroke with the onset 10-90 days prior to the enrollment
2. Age: 20-80y
3. With a hemiplegic upper extremity with Brunnstrom stage in I~IV
4. Able to understand simple orders (1-step orders, such as "raise your hand, touch your head….)
5. Totally independent in activity of daily life before the onset of stroke

Exclusion Criteria:

1. Incompliance to the assessments or interventions due to unstable medical condition, abnormal cognition, or other conditions.
2. Stroke of brainstem or cerebellum
3. Had received craniotomy or ventriculoperitoneal shunting
4. Needs of orthoses in walking before the onset of stroke
5. Had had motor dysfunctions (eg, amputation, cerebral palsy, poliomyelitis or other neuromuscular diseases) before the stroke.
6. Intracranial hemorrhage caused by artereovenous malformation, aneurysm, or tumor
7. Able to walk independently for more than 50 meters.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2020-05-20 (Estimated); Study Completion 2020-05-20 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment (upper extremity subscale) | 0-, 4- week
  The primary outcome is the change from baseline upper extremity subscale of Fugl-Meyer assessment at the end to 4-wk (post-intervention).

SECONDARY OUTCOMES:
Action Research Arm Test (ARAT) | 0-, 4-, 8-, 12-, 24 week
  A test that measures the upper extremity motor functions after the stroke.
Berg Balance Test | 0-, 4-, 8-, 12-, 24 week
  A test that measures the balance functions.
Fugl-Meyer Assessment (lower extremity subscale) | 0-, 4-, 8-, 12-, 24 week
  The FMA-LE (0-34) measures the lower extremity motor functions after the stroke.
Fugl-Meyer Assessment (upper extremity subscale) | 0-, 4-, 8-, 12-, 24 week
  FMA-UE (0-66), the subscale of FMA that measures the poststroke neuro-motor functions.
Time required for 10 meter walking | 0-, 4-, 8-, 12-, 24 week
  measuring the walking speed over a 10-meter distance
Stroke Impact Scale | 0-, 4-, 8-, 12-, 24 week
  A measure for stroke-specific quality of life
Barthel Index | 0-, 4-, 8-, 12-, 24 week
  to measure the activity of daily living

CONTACTS AND LOCATIONS:
Locations (1):
- WanFang Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Clark B, Whitall J, Kwakkel G, Mehrholz J, Ewings S, Burridge J. The effect of time spent in rehabilitation on activity limitation and impairment after stroke. Cochrane Database Syst Rev. 2021 Oct 25;10(10):CD012612. doi: 10.1002/14651858.CD012612.pub2. PMID 34695300